CLINICAL TRIAL: NCT03447561
Title: The Role of Consumption and Anticipation in Dopamine Release to Food Reward: an [18F]-Fallypride PET/MR Study.
Brief Title: The Role of Consumption and Anticipation in Dopamine Release to Food Reward
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Lukas Van Oudenhove, Associate Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: S60362-h
Record Dates: First submitted 2018-02-08; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Healthy; Food Reward
Keywords: Dopamine; Food; Reward; Anticipatory; Consummatory; Positron Emission Tomography; Magnetic Resonance; Metabolic hormones

STUDY DESIGN:
Intervention Model Description: All participants will receive one PETMR scan session with the combination of anticipatory (viewing high-calorie food images) and consummatory reward (drinking sips of chocolate milkshake), and one PETMR scan session with purely consummatory reward, in a randomized and counterbalanced order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anticipatory + consummatory food reward (Experimental): PET-MR scan session with a combination of anticipatory (viewing high-calorie food images) and consummatory food reward (drinking sips of chocolate milkshake). This scan session will consist of four blocks with a duration of 45 minutes each and 15 minute breaks in between. The first three blocks represent the 'control condition' (viewing neutral images and drinking sips of water) and the fourth block the 'food reward condition' (viewing high-calorie food images and drinking sips of chocolate milkshake).
  Interventions: Behavioral: Anticipatory + consummatory food reward
- Consummatory food reward (Experimental): PET-MR scan session with purely consummatory food reward (drinking sips of chocolate milkshake). This scan session will consist of four blocks with a duration of 45 minutes each and 15 minute breaks in between. The first three blocks represent the 'control condition' (drinking sips of water) and the fourth block the 'food reward condition' (drinking sips of chocolate milkshake).
  Interventions: Behavioral: Consummatory food reward

INTERVENTIONS:
Behavioral: Anticipatory + consummatory food reward — Exposure to a combination of anticipatory (viewing high-calorie food images) and consummatory food reward (drinking sips of chocolate milkshake).
  Arms: Anticipatory + consummatory food reward
Behavioral: Consummatory food reward — Exposure to consummatory food reward (drinking sips of chocolate milkshake).
  Arms: Consummatory food reward

SUMMARY:
This study aims to disentangle the relative contribution of the anticipatory (food images) versus consummatory (food administration) component of dopamine release to food reward, by performing simultaneous Positron Emission Tomography (PET) and Magnetic Resonance (MR) scanning. Additionally, this study aims to assess the relationship of the dopamine release with (changes in) metabolic hormone levels.

DETAILED DESCRIPTION:
The brain's reward system has a potent contribution to the regulation of food intake. Although animal work has demonstrated a key role of the mesolimbic dopamine system in food reward responses, evidence in humans is still sparse and inconsistent. Our research group recently used state-of-the-art Positron Emission Tomography (PET) imaging methods to study in vivo dopamine release in response to a combination of anticipatory (viewing high-calorie food images) and consummatory (drinking sips of chocolate milkshake) food stimuli in healthy women. The investigators demonstrated dopamine release in reward-related regions in the prefrontal cortex of the brain in response to these stimuli, correlating with levels of gastrointestinal hunger/satiety hormones, and predicting subsequent food intake.

The current study aims to disentangle the relative contribution of the anticipatory (food images) versus consummatory (food administration) component of dopamine release to food reward, by performing simultaneous Positron Emission Tomography (PET) and Magnetic Resonance (MR) scanning. Healthy females will participate in two PET-MR scan sessions in a fasted state: one session with the combination of anticipatory (viewing high-calorie food images) and consummatory reward (drinking sips of chocolate milkshake) and one session with purely consummatory reward. The order of these sessions will be randomized and counterbalanced.

Both scan sessions will consist of four blocks with a duration of 45 minutes each and 15 minute breaks in between. The first three blocks represent the 'control condition' and the fourth block the 'food reward condition'. At the end of each scan session, participants will take part in an ad libitum drink test in which they will be instructed to drink as much chocolate milkshake as preferred, until comfortably full. During both sessions, blood samples will be collected at several time points to assess levels of metabolic hormones and their relation to food-induced dopamine release. The proposed studies aims to increase our understanding of the psycho-biology of appetite and food intake regulation as well as identify potential new treatment targets for disorders of food intake, both at the level of the gastrointestinal tract and the brain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females (on hormonal contraception)
* Dutch-speaking
* Right-handed
* Stable body weight with Body Mass Index (BMI) of 18.5 - 25 kg/m^2

Exclusion Criteria:

* Medical, neurological or psychiatric disorders
* Use of psychotropic medication in past 6 months
* Use of cannabis or other drugs of abuse in past 12 months
* Lactose-intolerance or food allergies
* Vegetarian diet
* Smoking
* Consumption of more than 7 alcoholic units per week
* Exposure to a significant amount of ionizing radiation in past 12 months
* Claustrophobia
* Contra-indications for Magnetic Resonance Imaging
* Pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Dopamine release to combined vs consummatory food reward | Continuously over 225 minutes after onset scanning
  Changes in [18F]-Fallypride binding potential (reflecting dopamine release) in the food reward condition

SECONDARY OUTCOMES:
Composite measure of Metabolic hormone levels | 5 minutes before onset scanning and 45, 105, 165, 180, 195, 210 and 225 minutes after onset scanning
  Correlation between dopamine response to food reward and (changes in) metabolic hormone levels (ghrelin, motilin, glucagon-like peptide 1, peptide tyrosine tyrosine, leptin, and insulin).
Amount of milkshake consumed during drink test | 230 minutes after onset of scanning (immediately following end of scanning)
  Correlation between dopamine response to food reward and the amount of milkshake consumed during the drink test
Temperament and Character Inventory questionnaire | baseline, dopamine release measured 225 minutes following onset scanning
  Correlation between dopamine response to food reward and scores on the Temperament and Character Inventory questionnaire.

OTHER OUTCOMES:
Ratings of appetite-related sensations composite | 5 minutes before onset of scanning and several time-points up to 225 minutes after onset of scanning
  Ratings of hunger, fullness, prospective food consumption, satiety, nausea, pleasantness, liking, and wanting on Visual Analogue Scales

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Van Oudenhove, Prof. dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided